CLINICAL TRIAL: NCT04866641
Title: A Phase I, Open-label, Dose-finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of T-1201 Injection 100 mg Kit in Patients With Advanced Solid Tumors
Brief Title: Safety and Tolerability Study for T-1201 Injection 100 mg Kit in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taivex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAI-201
Record Dates: First submitted 2021-04-23; First posted 2021-04-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-1201 Injection 100 mg Kit (Experimental): T-1201 Injection 100 mg Kit will be administered via intravenous infusion once every 4 weeks (Part A), 2 weeks (Part B) or 3 weeks (Part C). T-1201 Injection 100 mg Kit is required to be reconstituted with its specific Injection Diluent supplied in the kit, then further diluted with 5% Dextrose solution prior to the intravenous infusion in patients.
  Interventions: Drug: T-1201 Injection 100 mg Kit

INTERVENTIONS:
Drug: T-1201 Injection 100 mg Kit — T-1201 Injection 100 mg Kit contains lyophilized powder with a sterile aqueous solution formulated for intravenous administration.

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of T-1201 injection in subjects with advanced solid tumors refractory to standard therapy, or for whom no standard therapy is available. The main questions it aims to answer are:

* The Maximum tolerated dose (MTD) of T-1201 on different dosing schedules.
* The Recommended Phase 2 dose (RP2D) of T-1201 on different dosing schedules.

Researchers will evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of T-1201.

Participants will:

Received T-1201 either once every 4 (Part A)/2 (Part B)/3 (Part C) weeks, depend on they participate in which parts of study.

Visit the clinic once every 2/3 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for enrollment in the study:

1. Signed and dated informed consent form.
2. Histologically and cytologically confirmed advanced malignancies that are refractory to standard therapy or have no accepted standard therapy.
3. Solid tumors that are measurable or evaluable as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion).
4. Female or male, 20 years of age or older.
5. ECOG performance status 0 or 1.
6. QTcF ≤ 470 ms at screening.

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

1. Clinically significant comorbidity such as unstable angina, congestive heart failure (NYHA Grade III or IV), uncontrolled hypertension (>160/100 mmHg despite optimal medical treatment), chronic obstructive pulmonary disease (COPD) with frequent exacerbations, refractory asthma, inflammatory bowel disease or intestinal obstruction.
2. Acute myocardial infarction or cerebrovascular accident (CVA) within 6 months prior the first dose of study drug.
3. Central nervous system (CNS) metastasis or seizure disorder due to underlying malignancy except those who have been treated and have stable CNS metastases or are asymptomatic.
4. AIDS-defining opportunistic infections within the past 12 months.
5. HBV infection (positive HBsAg) except for carrier of inactive HBV as defined by negative HBeAg with normal ALT and HBV DNA < 2,000 IU/mL or HCV infection (positive anti-HCV antibody) except for those with undetectable HCV RNA.
6. Inadequate bone marrow reserve, hepatic or renal function as defined by any of the following laboratory values:

   1. absolute neutrophil count (ANC) < 1500/µL
   2. platelet count < 100 x 10^9 /µL
   3. hemoglobin < 9 g/dL
   4. total bilirubin > 1.5 x the upper limit of normal (ULN)
   5. aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x ULN if no hepatic metastases are present; > 5 x ULN if hepatic metastases are present
   6. Estimated (Cockroft-Gault formula) creatinine clearance (CrCl) < 60 mL/min CrCl = [(140 - age (year)) x weight (kg)] / (serum creatinine x 72) (x 0.85 for females)
7. Toxicities resulting from prior therapy or surgical procedures not yet resolved to ≤ NCI CTCAE v5.0 Grade 1 with the exception of alopecia, skin hyperpigmentation or hypopigmentation.
8. Major surgical procedures (as defined by Investigator) within 4 weeks prior to the first dose of study drug or any ongoing post-operative complications.
9. Receiving any (investigational or approved) anti-cancer therapy (including chemotherapy or targeted therapy) within 28 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
10. A history of apparent allergic reactions to irinotecan, Tween 80 (dosed with prior treatment with prophylactic drug), and/or ethanol.
11. If female, is pregnant or breastfeeding.
12. If men or women with childbearing potential, unwilling to use effective contraceptive methods during the study and for at least 3 months (men) or 1 month (women) after the last dose of study drug. Effective contraceptive methods include implants, injectables, combined oral contraceptives, intra-uterine devices (IUDs), sexual abstinence, surgical sterilization or a partner who is sterile.
13. Receiving live attenuated vaccine within 28 days prior to the first dose of study drug.
14. Life expectancy < 3 months
15. Other prior or ongoing condition(s) that, in Investigator's opinion, could affect the safety of the subject, compromise the subject's ability to comply with the study requirements or impair the assessment of study results.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | First treatment cycle (i.e., the first 28 days post the first dose)
  MTD is highest dose level in which 6 patients have been treated with at most 1 experiencing dose limiting toxicity (DLT).
Recommended Phase 2 dose (RP2D) dose (RP2D) | First treatment cycle (i.e., the first 28 days post the first dose)
  To determine the recommended Phase 2 dose (RP2D)
Frequency, type, severity and relationship to study drug of adverse events (AEs) | At least 2 months
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
Pharmacokinetic profiles: Cmax of T-1201 and its metabolite(s) [0060 and SN-38] | 340 hours
  Maximum plasma concentration (Cmax ) of T-1201, 0060, and SN-38 from plasma concentration-time profiles.
Pharmacokinetic profiles: Tmax of T-1201 and its metabolite(s) [0060 and SN-38] | 340 hours
  Time to reach maximum concentration (Tmax ) of T-1201, 0060, and SN-38 from plasma concentration-time profiles.
Pharmacokinetic profiles: MRT of T-1201 and its metabolite(s) [0060 and SN-38] | 340 hours
  Mean residence time (MRT) of T-1201, 0060, and SN-38 from plasma concentration-time profiles.
Pharmacokinetic profiles: AUC of T-1201 and its metabolite(s) [0060 and SN-38] | 340 hours
  The area under the plasma concentration-time curve (AUC) of T-1201, 0060, and SN-38 from plasma concentration-time profiles.
Pharmacokinetic profiles: T1/2 of T-1201 and its metabolite(s) [0060 and SN-38] | 340 hours
  Terminal half-life (T1/2 ) of T-1201, 0060, and SN-38 from plasma concentration-time profiles.
Assess preliminary anti-tumor activity: ORR of T-1201 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | At least 56 days
  Objective response rate (ORR)
Assess preliminary anti-tumor activity: CBR of T-1201 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | At least 56 days
  Clinical benefit rate (CBR)
Assess preliminary anti-tumor activity: DOR of T-1201 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | At least 56 days
  Duration of response (DOR)
Assess preliminary anti-tumor activity of T-1201 according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | At least 56 days
  Time to tumor progression per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: Undecided